CLINICAL TRIAL: NCT05091762
Title: Effect of Physiological Ischemic Training on Patients With Atherosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, linaicui, Principal Investigator, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20210604-02
Record Dates: First submitted 2021-09-23; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Atherosclerosis
Keywords: resistance training
MeSH Terms: conditions — Atherosclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Blank control group (No Intervention)
- Exercise group (Experimental)
  Interventions: Behavioral: exercise
- Hyperlipidemia group (No Intervention)
- Hyperlipidemia and medication group (No Intervention)
- Hyperlipidemia and exercise group (Experimental)
  Interventions: Behavioral: exercise
- Hyperlipidemia and medication and exercise group (Experimental)
  Interventions: Behavioral: exercise
- Routine treatment group (No Intervention)
- Routine treatment and exercise group (Experimental)
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — Upper limb resistance training with blood flow obstruction
  Arms: Exercise group; Hyperlipidemia and exercise group; Hyperlipidemia and medication and exercise group; Routine treatment and exercise group

SUMMARY:
To study whether the resistance training with blood flow obstruction in patients in early atherosclerosis period can produce a beneficial effect on preventing atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. LDL > 3.11mmol/l and less than 5.63mmol/l;
2. No serious heart, blood vessel and other related diseases;
3. There were no skeletal and muscular diseases affecting sports training;
4. No regular exercise in the past half year (no more than 2 times a week, no more than 30 minutes each time);
5. Smoking less than 1 pack / year, no history of drinking.

Exclusion Criteria:

1. Haven't other serious heart and vascular diseases other than hyperlipidemia and / or bones and muscles that affect sports training Diseases;
2. Pregnant women and people with disabilities;
3. Other circumstances determined by the researcher not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endothelium dependent vasodilation | 8 weeks
  Percentage of the change
Blood lipid analysis results | 8 weeks
  Content of total cholesterol, triglycerides, high density lipoprotein and low density lipoprotein

SECONDARY OUTCOMES:
The inflammatory state | 8 weeks
  Content of NO, eNOS, iNOS, IFN-γ, IL-6, IL-10 in blood
Endothelial repair function | 8 weeks
  eNOSmRNA, iNOSmRNA, EPCs in blood

CONTACTS AND LOCATIONS:
Overall Officials: Aicui Lin, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No